CLINICAL TRIAL: NCT02254629
Title: The Effects of Laxative-probiotic Sequential Treatment on the Symptoms and Fecal Microbiota in the IBS Patients.
Brief Title: The Effects of Laxative-probiotic Sequential Treatment in the Irritable Bowel Syndrome Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014SDU-QILU-G04
Record Dates: First submitted 2014-08-28; First posted 2014-10-02 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: Fecal microflora; IBS; Sequential treatment; Probiotic; Laxative
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- laxative-probiotic sequential (Experimental): laxative：2000 ml. Probiotic：2 tablets/ times, 3 times / day for the first 2 weeks，immediately after colonoscopy
  Interventions: Drug: Probiotic Clostridium Butyricum; Drug: Laxative Polyethylene Glycol
- probiotic (Active Comparator): Probiotic：2 tablets/ times, 3 times / day for the first 2 weeks.
  Interventions: Drug: Probiotic Clostridium Butyricum
- Laxative followed by Probiotic 2 weeks later (Active Comparator): laxative：2000 ml. Probiotic：2 tablets/ times, 3 times / day for the last 2 weeks with two weeks interval after colonoscopy.
  Interventions: Drug: Probiotic Clostridium Butyricum; Drug: Laxative Polyethylene Glycol

INTERVENTIONS:
Drug: Probiotic Clostridium Butyricum — probiotic:2 tablets/ times, 3 times / day for 2 weeks
  Other Names: Clostridium Butyricum Tablets
Drug: Laxative Polyethylene Glycol — laxative：2000 ml.
  Other Names: Polyethylene Glycol Electrolytes Powder.
  Arms: Laxative followed by Probiotic 2 weeks later; laxative-probiotic sequential

SUMMARY:
the laxative-probiotic sequential treatment might reduce the symptoms of IBS and alter the fecal microbiota of the patients in a more robust manner .

DETAILED DESCRIPTION:
Probiotics can regulate intestinal immunity, repair mucosal barrier, and reportedly exert therapeutic effects on IBS patients. The laxatives could also alter the gut microflora significantly, thus the laxative-probiotic sequential treatment might affect the symptoms and the composition of fecal microbiota in the IBS patients in a more robust manner .

ELIGIBILITY:
Inclusion Criteria:

* the presence of Rome III criteria for IBS ;
* Patients scheduled for colonoscopy examination or having negative screening examinations
* Aged between 18 and 65 years old

Exclusion Criteria:

* Antibiotic, probiotic or laxative usage within 4 weeks.
* organic gastrointestinal diseases
* Severe systematic disease: diabetes mellitus, hepatic, renal or cardiac dysfunction, thyroid disease or tumor etc.
* pregnancy or lactation.
* previous major or complicated abdominal surgery.
* severe endometriosis and dementia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Subject's Global Assessment of Relief | 8 months
  The SGA (subjective global assessment) of Relief was assessed by answering the following question: "Please consider how you felt this past week in regard to your IBS, in particular your overall wellbeing, symptoms and altered bowel habit. Compared to the way you usually felt before entering the study, how would you rate your relief of symptoms during the past week?" The scale contained five possible answers: (1) completely relieved, (2) considerably relieved, (3) somewhat relieved, (4) unchanged, or (5) worse.

SECONDARY OUTCOMES:
The changes of symptom scores | 8 months
  The symptom score includes abdominal pain, discomfort, bloating, stool frequency, stool consistency according to Bristol stool form scale and defecation urgency，imcomplete，straining.
IBS patients'quality of life | 8 months
  Quality of life was determined by using IBS-QOL scoring system for patients with IBS. This questionnaire comprises a range of 34 items with response options on a 5-point rating scale. The items contribute to 8 domains as follows: Dysphoria, Interference with activity, Body image, Health worry, Food avoidance, Social reaction, Sexual, Relationship.
Composition of Microorganisms in stool | 8 months
  Primary coordination of fecal samples' 16s rDNA (ribosomal deoxyribonucleic acid) will be compared between two Groups using Braycurtis distance based Primary coordination analysis (PCoA).

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD.PhD, Principal Investigator — Qilu Hospital of Shandong University; Yanqing Li, MD.PhD., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Li M, Xu R, Li YQ. Sequential laxative-probiotic usage for treatment of irritable bowel syndrome: a novel method inspired by mathematical modelling of the microbiome. Sci Rep. 2020 Nov 9;10(1):19291. doi: 10.1038/s41598-020-75225-z. PMID 33168839